CLINICAL TRIAL: NCT05109988
Title: The Effect of a Father-involvement Breastfeeding Telephone Support Intervention on Exclusive and Sustained Breastfeeding: A Randomized Controlled Trial.
Brief Title: Father-involvement Telephone Support Intervention on Breastfeeding: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ngai Fei Wan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18191141
Record Dates: First submitted 2021-10-17; First posted 2021-11-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Feeding, Exclusive; Parents
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome measures will be collected by a research assistant who is blind to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of four weekly 20-30 minutes telephone-administered counselling sessions on breastfeeding, delivered individually in the first month postpartum for mothers and fathers.
  Interventions: Behavioral: Breastfeeding telephone support
- Control (No Intervention): Standard postpartum care

INTERVENTIONS:
Behavioral: Breastfeeding telephone support — The intervention consists of four weekly 20-30 minutes telephone-administered counselling sessions on breastfeeding, delivered individually in the first month postpartum for mothers and fathers.
  Arms: Intervention

SUMMARY:
The World Health Organization advocates for breastfeeding as the best source of food for optimal infant development, which reduces the risk of infant mortality and morbidity. The objectives of this study are to evaluate the effect of a father-involvement breastfeeding telephone support intervention on prevalence and duration of exclusive breastfeeding, postnatal depression and parent-infant bonding. The intervention consists of four weekly 20-30 minutes telephone-administered counselling sessions on breastfeeding, delivered individually in the first month postpartum for mothers and fathers. We expect that women who receive the intervention will have a higher rate and longer duration of exclusive breastfeeding, fewer depressive symptoms and better parent-child relationship. The knowledge gained from this study can provide direction for the development of flexible, accessible and culturally sensitive interventions to promote breastfeeding and mental health in Chinese society.

DETAILED DESCRIPTION:
Exclusive breastfeeding is recommended as the most beneficial form of infant nutrition during the first 6 months of life, which protects infants against childhood illness and reduces the risk of infant mortality and morbidity. The aim of this study is to implement and evaluate a breastfeeding telephone support intervention that involves mothers and fathers during the postpartum period. The objectives are to evaluate the effect of a father-involvement breastfeeding telephone support intervention on prevalence and duration of exclusive breastfeeding, postnatal depression and parent-infant bonding.

Hypothesis to be tested:

1. Mothers who receive the father-involvement telephone support intervention will have a higher rate and a longer duration of exclusive breastfeeding at 1, 2, 4 and 6 months postpartum than those who receive the standard postpartum care.
2. Mothers and fathers who receive the intervention will have: (a) fewer depressive symptoms, and (b) better parent-infant bonding at 2 and 6 months postpartum than those who receive the standard postpartum care.

Design and subjects: Randomized controlled trial. A sample of postpartum mothers (n = 738) and fathers (n = 738) will be randomly assigned to either the experimental or the control groups.

Study instruments: Edinburgh Postnatal Depression Scale (EPDS) and Postpartum Bonding Questionnaire (PBQ).

Intervention: The intervention consists of four weekly 20-30 minutes telephone-administered counselling sessions on breastfeeding, delivered individually in the first month postpartum for mothers and fathers.

Main outcome measures: The prevalence and duration of exclusive breastfeeding will be collected at 1, 2, 4 and 6 months postpartum. Postnatal depression and parent-infant boding will be assessed by the EPDS and the PBQ, respectively, at 2 and 6 months postpartum.

Data analysis: Generalized linear mixed models and survival analysis will be conducted to compare differences in the outcomes between two groups.

Potential application: The implementation of a simple, brief telephone-based intervention for breastfeeding families is most likely to be taken up in the primary health care setting. The results may better equip policy makers and health professionals to design health promotion programs for breastfeeding families, thus reducing the public health burden of childhood illness.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above;
* giving birth to a single healthy baby at term
* ability to speak and read the Chinese language

Exclusion Criteria:

* psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of exclusive breastfeeding | 1 month
  The prevalence/proportion of infants younger than 1 month who are exclusively breastfed is calculated as the number of infants younger than 1 month who are exclusively breastfed in the last 24 hours divided by the total number of infants younger than 1 month.

SECONDARY OUTCOMES:
Prevalence of exclusive breastfeeding | 2 months
  The prevalence of infants younger than 1 month who are exclusively breastfed is calculated as the number of infants younger than 1 month who are exclusively breastfed in the last 24 hours divided by the total number of infants younger than 1 month.
Prevalence of exclusive breastfeeding | 4 months
  The prevalence of infants younger than 4 months who are exclusively breastfed is calculated as the number of infants younger than 4 months who are exclusively breastfed in the last 24 hours divided by the total number of infants younger than 4 months.
Prevalence of exclusive breastfeeding | 6 months
  The prevalence of infants younger than 6 months who are exclusively breastfed is calculated as the number of infants younger than 6 months who are exclusively breastfed in the last 24 hours divided by the total number of infants younger than 6 months.
Duration of exclusive breastfeeding | 1 month
  The duration of exclusive breastfeeding is measured as the infant's age in weeks when the women first introduce infant formula.
Duration of exclusive breastfeeding | 2 months
  The duration of exclusive breastfeeding is measured as the infant's age in weeks when the women first introduce infant formula.
Duration of exclusive breastfeeding | 4 months
  The duration of exclusive breastfeeding is measured as the infant's age in weeks when the women first introduce infant formula.
Duration of exclusive breastfeeding | 6 months
  The duration of exclusive breastfeeding is measured as the infant's age in weeks when the women first introduce infant formula.
Edinburgh Postnatal Depression Scale | 2 months
  The Edinburgh Postnatal Depression Scale is a 10-item self-report instrument used to assess the presence of depressive symptoms during the postnatal period. Each item is scored on a 4-point scale and total scores ranging from 0 to 30, with higher scores indicating more depressive symptoms.
Edinburgh Postnatal Depression Scale | 6 months
  The Edinburgh Postnatal Depression Scale is a 10-item self-report instrument used to assess the presence of depressive symptoms during the postnatal period. Each item is scored on a 4-point scale and total scores ranging from 0 to 30, with higher scores indicating more depressive symptoms.
Postpartum Bonding Questionnaire | 2 months
  to assess parent-infant relationship
Postpartum Bonding Questionnaire | 6 months
  to assess parent-infant relationship

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wan Ngai, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ngai Fei Wan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No